CLINICAL TRIAL: NCT02241629
Title: Levo Phencynonate Hydrochloridefor the Prevention of Motion Sickness (Seasickness): a Randomized, Double-blind, Placebo Controlled, Multicenter,PhaseⅡClinical Study
Brief Title: Levo Phencynonate Hydrochloride for the Prevention of Seasickness
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sihuan Pharmaceutical Holdings Group Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: BOJI-1423Q
Record Dates: First submitted 2014-09-12; First posted 2014-09-16 (Estimated); Last update posted 2015-05-07 (Estimated); Status verified 2014-09

CONDITIONS: Motion Sickness
Keywords: motion sickness
MeSH Terms: conditions — Motion Sickness

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- levo phencynonate hydrochloride 1mg (Experimental): levo phencynonate hydrochloride tablet 1mg
  Interventions: Drug: placebo; Drug: levo phencynonate hydrochloride
- placebo (Placebo Comparator): Placebo
  Interventions: Drug: placebo
- levo phencynonate hydrochloride 2mg (Experimental): levo phencynonate hydrochloride 2mg
  Interventions: Drug: levo phencynonate hydrochloride

INTERVENTIONS:
Drug: placebo — placebo of levo phencynonate hydrochloride
  Arms: levo phencynonate hydrochloride 1mg; placebo
Drug: levo phencynonate hydrochloride — levo phencynonate hydrochloride
  Arms: levo phencynonate hydrochloride 1mg; levo phencynonate hydrochloride 2mg

SUMMARY:
A double-blind, randomized, placebo controlled, multicenter, dose-finding phaseⅡclinical superiority study.

DETAILED DESCRIPTION:
The trial is composed by 3 parts: 1) On-boat screening period for seasickness and safety tests will be evaluated in minus one day. 2) 4 weeks of washout period to eliminate the impact of voyage experience. 3) On-boat drug testing period. The subjects will be administered the drug before voyage. The seasickness symptoms will be evaluated during voyage. The safety test will be conducted before and after one day of on-boat testing.

ELIGIBILITY:
Inclusion Criteria:

* Subjects fulfilling the diagnostic criteria for motion sickness
* Have medical history for motion sickness
* During screening, the severity of sea sickness is assessed as moderate or above according to sea sickness severity scale.
* Adults for 18-55 years, male or female.
* Agree to participate the study and can sign the ICF independently.

Exclusion Criteria:

* Be allergic to the study drug or be allergic constitution
* ALT, AST≥ 1.5 times of ULN, Scr>ULN, or other clinical significant lab values.
* Abnormal ECG which is clinical significant judged by investigators, including: QTc>normal range
* Have medical history for urination disorder
* Have headache, vertigo, dizziness or nsomnia caused by other diseases than motion sickness.
* Have active gastrointestinal diseases or overweight (BMI≥24kg/m2 )
* Have internal ear disease which may disturb the evaluation of motion sickness.
* Have glaucoma or posterior circulation ischemia
* Have anxiety, depression or other mental disease that investigator considering inadaptable to participate the study.
* Participated in other studies within the past 3 months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 180 (Actual)
Dates: Start 2014-08; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
the symptoms of seasickness | Two hours of voyage
  Investigators should assess the symptoms of seasickness for subjects according to sea sickness severity scale.

CONTACTS AND LOCATIONS:
Overall Officials: Weiguo Xue, Principal Investigator — Qingdao Municipal Hospital
Locations (1):
- Qingdao municipal hospital, Qingdao, Shandong, China